CLINICAL TRIAL: NCT06678269
Title: A Phase I Study of Concurrent Abemaciclib and Radiation Therapy (RT) for Patients With Metastatic Hormone Receptor Positive (HR+), HER2 Negative (HER2-) Breast Cancer
Brief Title: A Study of Abemaciclib and Radiation Therapy in People With Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-138
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer; Stage IV Breast Cancer; Breast Cancer; Breast Cancer Stage IV; Breast Cancer Metastatic; HER2-negative Breast Cancer; HER2 Negative Breast Carcinoma; Hormone-receptor-positive Breast Cancer
Keywords: Metastatic Breast Cancer; Stage IV Breast Cancer; Breast Cancer; Breast Cancer Stage IV; Breast Cancer Metastatic; HER2-negative Breast Cancer; HER2 Negative Breast Carcinoma; Hormone-receptor-positive Breast Cancer; Memorial Sloan Kettering Cancer Center; 24-138
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with HR+, HER2- metastatic breast cancer (Experimental): Participants will have a diagnosis of HR+, HER2- metastatic breast cancer. Abemaciclib, orally every 12 (± 2) hours beginning on the day of simulation thru the final day of radiotherapy for a maximum 28-day course. Radiation therapy, 27Gy in 3 daily fractions or 30Gy in 5 daily fractions completed entirely within 28 days of simulation.
  Interventions: Drug: Abemaciclib; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Abemaciclib — The dose escalation portion of the study, a 3+3 design will be used. Once the MTD of Abemaciclib is reached, the phase Ib expansion portion will enroll up to 10 additional patients also requiring palliation to bone metastases
Radiation: Radiation Therapy — 27Gy in 3 daily fractions or 30Gy in 5 daily fractions completed entirely within 28 days of simulation via stereotactic body radiotherapy (SBRT).

SUMMARY:
The purpose of this study is to test different doses of abemaciclib to find the best dose in participants while receiving hormone therapy and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at signing of informed consent.
* Both male and female patients are allowed
* Histologically confirmed metastatic breast cancer (mBC), current stage IV.
* Plan for ablative radiotherapy (SBRT) to a bone metastasis.
* Documented estrogen receptor (ER) positive and/or progesterone receptor (PgR) positive by immunohistochemistry. The threshold to qualify as ER or PgR positive is ≥1% per ASCO/CAP guidelines.
* HER2 negative tumor status confirmed by immunohistochemistry or FISH per ASCO/CAP guidelines.
* Any line of prior treatments (hormonal therapy and chemotherapy) is permitted including prior abemaciclib, palbociclib and ribociclib.
* At the time of enrollment, treating physician has intent to resume abemaciclib (at any dose) following radiotherapy.
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment. A washout period of at least 21 days is required between last chemotherapy dose and enrollment (provided the patient did not receive radiotherapy).
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and enrollment. No prior radiotherapy to the current intended target site is permitted (ie. reirradiation is excluded from this study).
* The patient must be able to swallow oral medications.
* The patient must have adequate organ function per the following criteria (as defined in Table 2):

Table 2: Laboratory Value Guidance to Establish Adequate Organ Function Hematologic ANC: ≥1.5 x 10^9/L Platelets: ≥100 x 10^9/L Hemoglobin: ≥8 g/dL Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.

Hepatic Total bilirubin: ≤1.5 x ULN Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted ALT and AST: ≤3 x ULN

* Patient may remain on hormonal therapy and abemaciclib before enrollment.
* Patients must discontinue other CDK4/6 inhibitor (palbociclib or ribociclib) for at least 7 days and recover from the acute effects of therapy (until the toxicity resolves to ≤Grade 1) except for residual alopecia and peripheral neuropathy.
* Measurable or non-measurable disease is permitted as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
* Patients must have an Eastern Cooperative Oncology Group (ECOG) status of ≤2 or Karnofsky Performance Status (KPS) ≥60.
* Negative β-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause.
* Women of childbearing potential must agree and commit to the use of a highly effective method of contraception as determined to be acceptable by the investigator, from the time of informed consent until 28 days after the last dose of the investigational product. Men must agree and commit to use a barrier method of contraception while on treatment and for 4 weeks after last dose of investigational products.
* Patients (or their legally authorized representative) must provide written, informed consent to participate in the study and follow the study procedures
* At the discretion of the treating radiation oncologist, radiation to a metastatic bone lesion is indicated inclusive of bone lesions in the spinal column.

Exclusion Criteria:

* Bone lesions in the calvarium are not eligible for the dose-finding or expansion portions of the study.
* Patients currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* The patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to the start of study intervention, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.
* Patients who received radiation therapy ≤14 days prior to initiation of investigational agents are excluded.
* Patients are ineligible if they have serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Females who are pregnant or lactating.
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade ≥2 diarrhea of any etiology screening).
* Malignant spinal cord compression (ESCC2 or above)
* Prior radiation therapy to the current target site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/MTD of abemaciclib | up to 1 year
  The primary endpoint of the study is defining the MTD of abemaciclib in combination with Radiation Therapy/RT

CONTACTS AND LOCATIONS:
Overall Officials: Lior Braunstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org